CLINICAL TRIAL: NCT00102206
Title: A Phase II, Randomized, Open-Label Study to Evaluate the Safety and Effectiveness of Two Antiretroviral Therapeutic Strategies: A Dual PI-Based HAART Regimen Versus a Multi-NRTI ART Regimen, in ART-Experienced Children and Youth Who Have Experienced Virologic Failure
Brief Title: A Comparison of Two Anti-HIV Drug Regimens for Youth Who Have Failed Prior Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1053; 10131 (Registry Identifier: DAIDS ES); PACTG P1053
Record Dates: First submitted 2005-01-25; First posted 2005-01-26 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Child
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Emtricitabine; Lamivudine; Lopinavir; Saquinavir; Tenofovir; Zidovudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Emtricitabine
Drug: Lamivudine
Drug: Lopinavir/ritonavir
Drug: Saquinavir
Drug: Tenofovir disoproxil fumarate
Drug: Zidovudine

SUMMARY:
HIV infected children and adolescents who have taken many anti-HIV drugs may have limited treatment options and are at high risk for progressing to AIDS. The purpose of this study is to determine whether an anti-HIV treatment regimen of 2 protease inhibitors (PIs) and 2 nucleoside reverse transcriptase inhibitors (NRTIs) is more effective than a regimen of 4 NRTIs in treatment-experienced children and adolescents who have failed previous anti-HIV treatment.

DETAILED DESCRIPTION:
HIV infected children and adolescents on anti-HIV treatment regimens have traditionally had more difficulty with non-adherence and drug resistance than adults, often resulting in virologic failure. Additionally, HIV infected children with extensive exposure to antiretrovirals (ARVs) are likely to have fewer therapeutic options for salvage therapy, and their physicians find it difficult to choose regimens that will keep the HIV infection under control. This study will compare the efficacy of three 4-drug ARV salvage regimens in treatment-experienced, HIV infected children and adolescents who have experienced virologic failure.

This study will last at least 96 weeks. Participants will be randomly assigned to one of three groups. Group 1A will receive a dual-PI based regimen of lopinavir/ritonavir (LPV/r), saquinavir (SQV), and the NRTIs emtricitabine (FTC) and abacavir sulfate (ABC). Group 1B will receive a dual-PI based regimen of LPV/r, SQV, FTC, and tenofovir disoproxil fumarate (TDF). Group 2 will receive an NRTI-only regimen of ABC, lamivudine, zidovudine, and TDF.

There will be 11 study visits during Step I of this study. Medical history, a physical exam, and blood collection will occur at all visits. Dual-energy x-ray absorptiometry (DEXA) scans will occur at study entry and at Weeks 24, 48, 72, and 96. Urine collection will occur at most visits; participants will also take part in adherence modules at most visits. Participants will be asked to complete a pill count form at Weeks 4 and 24. Additionally, some study participants will be asked to participate in an intensive pharmacokinetics study at Week 4.

ELIGIBILITY:
Inclusion Criteria for Step I:

* HIV infected
* No currently available therapeutic options that would likely result in long-term suppression of virus to less than 400 copies/ml
* Two measurements within 4 months prior to screening and at screening of either CD4% of less than 15% and HIV viral load of greater than 10,000 copies/ml OR HIV viral load greater than 30,000 copies/ml
* Previous exposure to non-nucleoside reverse transcriptase inhibitors (NNRTIs), NRTIs, and PIs AND have experienced virologic failure. More information on previous treatment regimen requirements is available in the protocol.
* Prior or current virologic failure with genotypic or phenotypic resistance OR historical virologic failure with a PI- or NNRTI-containing regimen
* Resistance to 2 or more drugs in most recent treatment regimen within 26 weeks prior to study screening
* Able and willing to swallow study medications
* Parent or guardian willing to provide informed consent, if applicable
* Willing to use acceptable methods of contraception

Exclusion Criteria for Step I:

* Previous cumulative exposure to TDF for more than 24 weeks OR more than 14 days of TDF exposure during the 24 weeks prior to study entry
* Grade 1 lipase or higher within 28 days prior to study entry
* Grade 3 or higher laboratory abnormality (except for lipase) within 28 days prior to study entry
* History of allergy or hypersensitivity to any of the study drugs
* Active CDC Stage C opportunistic infection or serious bacterial infection requiring therapy at the time of screening
* Chemotherapy for active cancer
* Require certain medications
* Abnormal kidney function
* Any clinically significant diseases other than HIV infection or findings during medical history screening that, in the opinion of the investigator, may interfere with the study
* Pregnancy or breastfeeding

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Tolerability of dual PI-based HAART versus multi-NRTI HAART salvage regimens (time to first intolerant event)
95% confidence interval (CI) for change in CD4% computed for PI-containing groups versus PI-sparing group
95% CI for change in BMD (both percent change in BMD and change in z-score from baseline) for each treatment group

SECONDARY OUTCOMES:
HIV-1 RNA
growth and development markers
toxicity
adherence
pharmacokinetics
special virologic and immunologic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wiznia, MD, Study Chair — Jacobi Medical Center; Ann J. Melvin, MD, MPH, Study Chair — Seattle Children's Hospital and Regional Medical Center
Locations (4):
- United States (4):
  - Chicago Children's CRS, Chicago, Illinois
  - Columbia IMPAACT CRS, New York, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - DUMC Ped. CRS, Durham, North Carolina

REFERENCES:
- [Background] Brogly S, Williams P, Seage GR 3rd, Oleske JM, Van Dyke R, McIntosh K; PACTG 219C Team. Antiretroviral treatment in pediatric HIV infection in the United States: from clinical trials to clinical practice. JAMA. 2005 May 11;293(18):2213-20. doi: 10.1001/jama.293.18.2213. PMID 15886376
- [Background] Gavin PJ, Yogev R. The role of protease inhibitor therapy in children with HIV infection. Paediatr Drugs. 2002;4(9):581-607. doi: 10.2165/00128072-200204090-00004. PMID 12175273
- [Background] Handforth J, Sharland M. Triple nucleoside reverse transcriptase inhibitor therapy in children. Paediatr Drugs. 2004;6(3):147-59. doi: 10.2165/00148581-200406030-00002. PMID 15170362
- [Background] Neely M, Kovacs A. Management of Antiretroviral Therapy in Neonates, Children, and Adolescents. Curr Infect Dis Rep. 2003 Dec;5(6):521-530. doi: 10.1007/s11908-003-0097-4. PMID 14642195
- [Background] Piketty C, Race E, Castiel P, Belec L, Peytavin G, Si-Mohamed A, Gonzalez-Canali G, Weiss L, Clavel F, Kazatchkine MD. Efficacy of a five-drug combination including ritonavir, saquinavir and efavirenz in patients who failed on a conventional triple-drug regimen: phenotypic resistance to protease inhibitors predicts outcome of therapy. AIDS. 1999 Jul 30;13(11):F71-7. doi: 10.1097/00002030-199907300-00001. PMID 10449277